CLINICAL TRIAL: NCT01253863
Title: Study of Accuracy of Preoperative Examination in Penetrating Wound
Brief Title: Diagnostic Accuracy of the Preoperative Clinical Examination in Upper Limb Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy/Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASD-1213-7
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2006-08

CONDITIONS: Penetrating Injury in Upper Limb
Keywords: Clinical Examination, Accuracy, Hand, Tendon, Injury.
MeSH Terms: conditions — Wounds and Injuries | interventions — Space Flight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- determining damaged tissue (Other)
  Interventions: Other: exploration

INTERVENTIONS:
Other: exploration — exploration of wound for determining damaged tissue

SUMMARY:
The purpose of this study is to determine the accuracy of preoperative clinical examination in penetrating injuries

DETAILED DESCRIPTION:
Penetrating injuries is a common cause of severe neurovascular damage, both in adults and children.we evaluated the accuracy of the preoperative clinical examination in depicting lesions caused by penetrating wounds of hands or forearms.

ELIGIBILITY:
Inclusion Criteria:

Deep penetrating injury to upper limb

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
number of determined tendon | 5 min after admission
  we evalauted tendon injuries without exploration of wound

SECONDARY OUTCOMES:
number of determined injured nerves | 5 min after admision
  we evaluated the number of detemined injured nerves without exploration of wound
number of damaged arteries | 5 min after admission
  we evaluated the number of detemined injured arteries without exploration of wound

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran